CLINICAL TRIAL: NCT00330408
Title: Impact of Training of GPs on Adherence of Hypertensive Individuals to Antihypertensive Medication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aga Khan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 05GS002MSC
Record Dates: First submitted 2006-05-25; First posted 2006-05-26 (Estimated); Last update posted 2006-05-26 (Estimated); Status verified 2006-04

CONDITIONS: Hypertension
Keywords: Adherence; GP training; Medication Event Monitoring System(MEMS); Antihypertensive Medication; Hypertension
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Behavioral: GP training

SUMMARY:
This study aims to assess the impact of training General Practitioners (GPs) on adherence to antihypertensive medication among hypertensive individuals. It also aims to assess risk factors for non-adherence. Special training (in appropriate algorithms for management and patient involvement in therapeutic decision making) has been given to GPs. The study has been conducted in six middle or low income clusters of Karachi recruiting individuals randomized to specially trained or untrained GPs, with a follow-up period of 6 weeks. The medication event monitoring system (MEMS)has been used for assessing adherence. It is hypothesized that compliance levels of individuals going to specially trained GPs is higher compared to those going to GPs not having received special training.

DETAILED DESCRIPTION:
Background: Lack of medication compliance is reported as a major factor contributing to inadequate control over blood pressure. Data from well-structured and well-conducted researches in this field, specifically in the context of developing countries is lacking.

Rationale: Targeting factors associated with non-adherence identified in this study would lead to reduction of the burden of poorly controlled hypertension and its complications. The special training of GPs, taken as an intervention in this study, if found successful in improving compliance, would be advocated for inclusion in a nation-wide hypertension control program.

Aims:

1. To assess difference in adherence to antihypertensive medication among hypertensive individuals visiting specially trained GPs, versus those visiting untrained GPs.
2. To assess risk factors associated with non-adherence

Study Design: Randomised Controlled Trial

Parent Study: This project stems from the population-based parent study "Population based strategies for effective control of high blood pressure in Pakistan"; a factorial design study. It is being conducted in twelve middle to low socioeconomic clusters of Karachi. These clusters are randomised to care by specially trained general practitioners (GP) vs. untrained GPs. Special training of GPs include rigorously training in appropriate algorithms for management, and patient involvement in therapeutic decision making.

Methodology: The target population for this study has been drawn from the parent study. 6 clusters randomized to the GP training intervention were selected. The specially trained GPs from the parent study are the intervention in this research. Hypertensive individuals from within the chosen clusters have been randomly selected for enrollment in the study. Patients going to specially trained or untrained GPs were taken as exposed or unexposed to the intervention, and were followed up for a month and a half months, in order to assess their adherence to antihypertensive medication. Adherence was further assessed with the help of the Medication Event Monitoring System (MEMS), which gives the date and time of when each bottle was opened. this method does not however ensure ingestion of the drug.

Intervention: GPs trained in appropriate algorithms for management and patient involvement in therapeutic decision making

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive individuals aged 40 years and above residing in selected clusters
* Individuals prescribed with hypertensive medication by their general practitioners in related cluster

Exclusion Criteria:

* Pregnant women will be excluded
* Mentally unstable or bed bound patients

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178
Dates: Start 2005-09; Study Completion 2006-04

PRIMARY OUTCOMES:
adherence:% of days correct dose was taken

SECONDARY OUTCOMES:
adherence: % prescribed doses taken

CONTACTS AND LOCATIONS:
Overall Officials: Tazeen H Jafar, MD, MPH, Study Director — Aga Khan Univeristy; Nudrat Qureshi, MSc Genetics, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Qureshi NN, Hatcher J, Chaturvedi N, Jafar TH; Hypertension Research Group. Effect of general practitioner education on adherence to antihypertensive drugs: cluster randomised controlled trial. BMJ. 2007 Nov 17;335(7628):1030. doi: 10.1136/bmj.39360.617986.AE. Epub 2007 Nov 8. PMID 17991935